CLINICAL TRIAL: NCT00419562
Title: Oral Insulin for Prevention of Diabetes in Relatives at Risk for Type 1 Diabetes Mellitus
Acronym: TN07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Center for Research Resources (NCRR) (NIH); American Diabetes Association (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TN07 Oral Insulin; UC4DK106993 (NIH); UC4DK117009 (NIH)
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: oral insulin; autoantigen; self tolerance; oral tolerance; Diabetes Prevention Trial - 1 (DPT-1); prevention; "at risk" for developing type 1 diabetes; juvenile diabetes; Type 1 diabetes (T1D); diabetes mellitus; Type 1 diabetes TrialNet; TrialNet
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Insulin (Experimental): 7.5 mg oral insulin capsules given before breakfast on a daily basis.
  Interventions: Drug: Oral Insulin
- Placebo (Placebo Comparator): Placebo capsule designed to match appearance of treatment capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Insulin — 7.5 mg oral insulin or placebo given before breakfast on a daily basis.
  Arms: Oral Insulin
Drug: Placebo — Placebo capsule designed to match active drug
  Arms: Placebo

SUMMARY:
Type 1 diabetes (T1D) is an autoimmune disease. This means that the immune system (the part of the body which helps fight infections) mistakenly attacks and destroys the cells that produce insulin (islet cells found in the pancreas). As these cells are destroyed, the body's ability to produce insulin decreases. There is evidence suggesting that repeated oral administration of an autoantigen (the same protein that the immune system is reacting to) may introduce a protective immunity and cause the immune system to stop its attack. An earlier, large scale study was done to see if oral insulin could delay or prevent the development of Type 1 diabetes in relatives at risk for developing Type 1 diabetes. The overall results showed that for the entire study population, oral insulin did not delay or prevent Type 1 diabetes. However, an analysis that was done after the conclusion of the trial suggested a potential beneficial effect in a subgroup of participants. The participants who seemed to benefit from oral insulin had higher levels of insulin autoantibodies which are directed against insulin itself ( called mIAA).

The Type 1 Diabetes TrialNet study group will further explore the potential role of oral insulin to delay or prevent Type 1 diabetes in a similar group of people. The study will also include a secondary group of individuals at different levels of risk than those in the primary cohort to gather information for future studies.

DETAILED DESCRIPTION:
Eligible participants will be randomized to receive either oral insulin (7.5 mg of recombinant human insulin crystals) or placebo daily.

All participants randomized into this study will be seen at a study site for a follow-up evaluation, three and six months after randomization, and every six months thereafter. Participants will be contacted by phone between 6-monthly clinic visits to assess changes in diabetes status, medication compliance and adverse events. These phone contacts will occur approximately 3 months from the date of the participants previous clinic visit.

At the study visits, participants will undergo assessments of their insulin production, immunologic status, and overall health. As the primary outcome measure, subjects will be followed until development of type 1 diabetes or the conclusion of the study. The trial is expected to last approximately 7-8 years or until the required amount of information is gathered.

ELIGIBILITY:
Inclusion Criteria:

1. Have a proband with Type 1 diabetes mellitus (T1DM). A proband is an individual diagnosed with diabetes before age 40 and started on insulin therapy within 1-year of diagnosis. Probands considered to have type 1 diabetes by their physician who do not meet this definition will be referred to the TrialNet Eligibility Committee.
2. If the proband is a parent, sibling or a child, the study participant must be 3 -45 years of age. If the proband is a second or third degree relative (i.e. niece, nephew, aunt, uncle, grandparent, cousin, or half-sibling), the study participant must be 3-20 years of age.
3. Willing to sign Informed Consent Form.
4. Oral glucose tolerance test (OGTT) performed within 7 weeks prior to randomization in which:

   * fasting plasma glucose < 110 mg/dL (6.1 mmol/l), and
   * 2 hour plasma glucose < 140 mg/dL (7.8 mmol/l)
5. mIAA confirmed positive within the previous six months.
6. Two samples with at least one autoantibody other than mIAA positive within the previous six months.

Exclusion Criteria:

1. Does not satisfy the above inclusion criteria. Subjects with mIAA positive but no other autoantibodies positive are not eligible for randomization.
2. Has severe active disease, e.g. chronic active hepatitis, severe cardiac, pulmonary, renal, hepatic, immune deficiency and/or disease that is likely to limit life expectancy or lead to therapies such as immunosuppression during the time of the study.
3. Prior participation in a trial for prevention of T1DM, e.g. nicotinamide, insulin, immunosuppressive drugs.
4. History of treatment with insulin or oral hypoglycemic agent.
5. History of therapy with immunosuppressive drugs or glucocorticoids within the past two years for a period of more than three months.
6. Ongoing use of medications known to influence glucose, i.e. sulfonylureas, growth hormone, metformin, anticonvulsants, thiazide or potassium depleting diuretics, beta adrenergic blockers, niacin. Subjects on such medications should be changed to a suitable alternative, if available, and will become eligible one month after medication is discontinued.
7. Pregnant or intends to become pregnant while on study or lactating.
8. Deemed unlikely or unable to comply with the protocol.
9. OGTT that reveals Diabetes, Impaired Glucose Tolerance (IGT), or Impaired Fasting Glucose (IFG).

   Diabetes is defined by:
   * fasting plasma glucose ³ 126 mg/dL (7 mmol/l), OR
   * 2 hour plasma glucose ³ 200 mg/dL (11.1 mmol/l)

   IGT is defined by:
   * fasting plasma glucose < 126 mg/dL (7 mmol/l), and
   * 2 hour plasma glucose 140-199 mg/dL (7.8 - 11mmol/l),

   IFG is defined by:
   * fasting plasma glucose 110-125 mg/dL (6.1-6.9 mmol/l) AND
   * 2 hour plasma glucose < 140 mg/dL (7.8 mmol/l)
10. Subject has HLA DQA1*0102, DQB1*0602 haplotype.

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 560 (Actual)
Dates: Start 2007-02; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Greenbaum, M.D., Study Chair — Benaroya Research Institute; Jeff Krischer, Ph.D., Principal Investigator — University of South Florida
Locations (18):
- United States (13):
  - University of California-San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Eskind Diabetes Clinic, Nashville, Tennessee
  - University of Texas, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Walter and Eliza Hall Institute, Parkville, Victoria, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- University of Turku, Turku, Finland
- San Raffaele Hospital, Milan, Italy
- University of Bristol, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/tn07-oral-insulin/?query=tn07
URL: https://repository.niddk.nih.gov/studies/tn07-oral-insulin/?query=tn07

REFERENCES:
- [Background] Bergerot I, Fabien N, Maguer V, Thivolet C. Oral administration of human insulin to NOD mice generates CD4+ T cells that suppress adoptive transfer of diabetes. J Autoimmun. 1994 Oct;7(5):655-63. doi: 10.1006/jaut.1994.1050. PMID 7840857
- [Background] Muir A, Schatz D, Maclaren N. Antigen-specific immunotherapy: oral tolerance and subcutaneous immunization in the treatment of insulin-dependent diabetes. Diabetes Metab Rev. 1993 Dec;9(4):279-87. doi: 10.1002/dmr.5610090408. No abstract available. PMID 7924825
- [Background] Muir A, Peck A, Clare-Salzler M, Song YH, Cornelius J, Luchetta R, Krischer J, Maclaren N. Insulin immunization of nonobese diabetic mice induces a protective insulitis characterized by diminished intraislet interferon-gamma transcription. J Clin Invest. 1995 Feb;95(2):628-34. doi: 10.1172/JCI117707. PMID 7860747
- [Background] Zhang ZJ, Davidson L, Eisenbarth G, Weiner HL. Suppression of diabetes in nonobese diabetic mice by oral administration of porcine insulin. Proc Natl Acad Sci U S A. 1991 Nov 15;88(22):10252-6. doi: 10.1073/pnas.88.22.10252. PMID 1946445
- [Background] Skyler JS, Krischer JP, Wolfsdorf J, Cowie C, Palmer JP, Greenbaum C, Cuthbertson D, Rafkin-Mervis LE, Chase HP, Leschek E. Effects of oral insulin in relatives of patients with type 1 diabetes: The Diabetes Prevention Trial--Type 1. Diabetes Care. 2005 May;28(5):1068-76. doi: 10.2337/diacare.28.5.1068. PMID 15855569
- [Background] Lachin JM. Maximum information designs. Clin Trials. 2005;2(5):453-64. doi: 10.1191/1740774505cn115oa. PMID 16315649
- [Result] Writing Committee for the Type 1 Diabetes TrialNet Oral Insulin Study Group; Krischer JP, Schatz DA, Bundy B, Skyler JS, Greenbaum CJ. Effect of Oral Insulin on Prevention of Diabetes in Relatives of Patients With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2017 Nov 21;318(19):1891-1902. doi: 10.1001/jama.2017.17070. PMID 29164254
- See also: Type 1 Diabetes TrialNet — http://www.diabetestrialnet.org
- See also: American Diabetes Association — http://www.diabetes.org
- See also: Juvenile Diabetes Foundation International — http://www.jdrf.org

RESULTS

PARTICIPANT FLOW:
Groups:
- 7.5 mg Oral Insulin Capsules: given before breakfast on a daily basis.
- Placebo Capsule: designed to mimic appearance of treatment capsule
Period: Overall Study
Arm/Group | 7.5 mg Oral Insulin Capsules | Placebo Capsule
Started | 283 | 277
Completed | 250 | 246
Not Completed | 33 | 31
Not completed — Lost to Follow-up | 12 | 13
Not completed — Withdrawal by Subject | 20 | 18
Not completed — Participant Institutionalized | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo capsule designed to mimic appearance of treatment capsule
- Total: Total of all reporting groups
Arm/Group | Oral Insulin | Placebo | Total
Number analyzed (Participants) | 283 | 277 | 560
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8.2 [5.9 to 12.5] | 8.2 [5.4 to 11.5] | 8.2 [5.7 to 12.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 107 | 220
  Male | 170 | 170 | 340
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 25 | 52
  Not Hispanic or Latino | 256 | 252 | 508
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was collected based on self-report
  Participants
    Self-Reported Race: White | 252 | 249 | 501
    Self-Reported Race: African American | 8 | 9 | 17
    Self-Reported Race: Asian/Pacific Islander | 4 | 6 | 10
    Self-Reported Race: Not Reported | 19 | 13 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 17 | 15 | 32
  United States | 226 | 227 | 453
  Finland | 4 | 5 | 9
  Italy | 7 | 7 | 14
  United Kingdom | 6 | 6 | 12
  Australia | 7 | 4 | 11
  Sweden | 5 | 3 | 8
  Germany | 9 | 6 | 15
  New Zealand | 3 | 5 | 8
Stratum [Count of Participants; unit: Participants] — 4 stratum defined by autoantibodies & beta cell functioning; autoantibodies include: microinsulin autoantibody (mIAA), islet cell autoantibodies (ICA), insulinoma associated antigen-2 (ICA512), & glutamic acid decarboxylase (GAD65)
  1. Positive for mIAA & positive for either ICA or ICA512 & GAD65; high functioning beta cells (primary)
  2. Positive for mIAA & positive for either ICA or ICA512 & GAD65; low functioning beta cells
  3. Positive for mIAA & positive for ICA512 or GAD65; high functioning beta cells
  4. Positive for mIAA & positive for ICA512 or GAD65; low functioning beta cells
  Participants
    1 | 203 | 186 | 389
    2 | 28 | 27 | 55
    3 | 51 | 63 | 114
    4 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Type 1 Diabetes Per Year Among Individuals in the Primary Stratum When Treated With Oral Inulin Versus Placebo
Description: Primary outcome is reported as the rate of type 1 diabetes per year among the primary stratum; type 1 diabetes was diagnosed based on metabolic testing and assessment of symptoms. This is calculated by dividing the number of participants who develop diabetes by the total number of years of follow-up.
Time Frame: Metabolic and immunological tests were conducted every 6 months; participants were followed for a median of 2.7 years
Measure: Number (95% Confidence Interval); unit: Proportion with diabetes/year
Arm/Group | Oral Insulin | Placebo
Number analyzed (Participants) | 203 | 186
Proportion with diabetes/year | 0.088 [0.067 to 0.112] | 0.102 [0.078 to 0.129]

2. Secondary Outcome: Rate of Type 1 Diabetes Per Year in Secondary Stratum (Stratum 2) When Treated With Oral Insulin Versus Placebo
Description: Secondary outcome is reported as the rate of type 1 diabetes per year among secondary stratum 2; type 1 diabetes was diagnosed based on metabolic testing and assessment of symptoms. This is calculated by dividing the number of participants who develop diabetes by the total number of years of follow-up.
Time Frame: Metabolic and immunological tests were conducted every 6 months; participants were followed for a median of 2.7 years
Population: Stratum 2: mIAA Confirmed, (ICA Confirmed) OR (ICA Not Confirmed AND ICA512+ AND GAD65ab+), low functioning beta cells
Measure: Number (95% Confidence Interval); unit: Proportion with diabetes/year
Arm/Group | Oral Insulin | Placebo
Number analyzed (Participants) | 28 | 27
Proportion with diabetes/year | 0.181 [0.096 to 0.291] | 0.341 [0.206 to 0.511]

3. Secondary Outcome: Rate of Type 1 Diabetes in Secondary Stratum (Stratum 3+4) When Treated With Oral Insulin Versus Placebo
Description: Secondary outcome is reported as the rate of type 1 diabetes per year among secondary stratum 3+4; type 1 diabetes was diagnosed based on metabolic testing and assessment of symptoms. This is calculated by dividing the number of participants who develop diabetes by the total number of years of follow-up.
Time Frame: Metabolic and immunological tests were conducted every 6 months; participants were followed for a median of 2.7 years
Population: Combine stratum 3 (mIAA Confirmed, ICA Not Confirmed, ICA512+ OR GAD65ab+, high functioning beta cells) and stratum 4 (mIAA Confirmed, ICA Not Confirmed, ICA512+ OR GAD65ab+, low functioning beta cells)
Measure: Number (95% Confidence Interval); unit: Proportion with diabetes/year
Arm/Group | Oral Insulin | Placebo
Number analyzed (Participants) | 52 | 64
Proportion with diabetes/year | 0.051 [0.026 to 0.086] | 0.047 [0.022 to 0.080]

ADVERSE EVENTS:
Arm/Group | Oral Insulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/283 | 0/277
Serious Adverse Events (participants affected / at risk) | 0/283 | 0/277
Other Adverse Events (participants affected / at risk) | 150/283 | 133/277
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Insulin (N=283) | Placebo (N=277)
Infection (Infections and infestations) | 67 (134) | 62 (120)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 30 (51) | 30 (37)
Endocrine (Endocrine disorders) | 18 (18) | 12 (12)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 38 (45) | 18 (20)
Allergy/Immunology (Immune system disorders) | 17 (18) | 11 (11)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 25 (29) | 18 (20)
Gastrointestinal (Gastrointestinal disorders) | 28 (30) | 25 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No